CLINICAL TRIAL: NCT04829916
Title: A Phase 1b, Randomised, Double-Blind, Parallel Treatment Group Clinical Study to Evaluate the Safety, Tolerability and Pharmacokinetics of RMC-035 in Subjects Undergoing Non-Emergent On-Pump Coronary Artery Bypass Graft and/or Valve Surgery
Brief Title: A Study to Evaluate RMC-035 in Subjects Undergoing Cardiac Surgery
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Guard Therapeutics AB (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20-ROS-04
Record Dates: First submitted 2021-03-26; First posted 2021-04-02 (Actual); Results first posted 2023-12-04 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Acute Kidney Injury (AKI)
Keywords: AKI
MeSH Terms: conditions — Acute Kidney Injury | interventions — Solutions; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RMC-035 (Experimental): Participants will receive RMC-035 intravenously
  Interventions: Drug: RMC-035
- Placebo (Placebo Comparator): Participants will receive matching placebo solution intravenously
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RMC-035 — Multiple dosing during 48 hours following cardiac surgery
  Other Names: Solution for injection
  Arms: RMC-035
Drug: Placebo — Multiple dosing during 48 hours following cardiac surgery
  Other Names: Solution for injection
  Arms: Placebo

SUMMARY:
The purpose of the clinical study is to assess safety, tolerability and pharmacokinetics of RMC-035 for the prevention and treatment of acute kidney injury (AKI) in patients undergoing cardiac surgery.

DETAILED DESCRIPTION:
This is a study with two parallel treatment groups where subjects are randomized to receive RMC-035 or a matching placebo in a double-blind fashion. The study will comprise of a screening visit, followed by CABG and/or valve replacement on Day 1, double-blind treatment period and a follow-up period up to Day 30.

ELIGIBILITY:
Key Inclusion Criteria:

* Female and male subjects with an age ≥18 years
* Subject is scheduled for non-emergent (elective) CABG and/or valve surgery (single or multiple valves) with use of cardiopulmonary bypass (CPB)
* Subject has at least ONE of the following risk factors for AKI at screening:

  * History of LVEF <35% for at least 3 months prior to screening assessed by either echocardiography, cardiac MRI or nuclear scan.
  * History of previous open chest cavity cardiac surgery with or without CPB
  * Confirmed diagnosis of type 2 diabetes (T2DM) at least 3 months prior to screening AND ongoing treatment with an approved anti-diabetic drug
  * Age ≥70 years
  * Documented history of heart failure NYHA class II or higher for at least 3 months or longer at screening
  * Documented history of previous AKI before date of screening independent of the etiology of AKI
  * Documented history of anemia with hemoglobin ≤ 11 g/dL (≤6.8 mmol/L) for at least 3 months prior to screening
  * Documented history of albuminuria, defined as UACR >30 mg/g or > 30 mg/24 hour in a 24-hour urine collection.
  * eGFR is ≤ 60 mL/min/1.73 m2 using the Chronic Kidney Disease - Epidemiology Collaboration (CKD-EPI) equation

Key Exclusion Criteria:

* Estimated glomerular filtration rate (eGFR) is <30 mL/min/1.73 m2 using the Chronic Kidney Disease - Epidemiology Collaboration (CKD-EPI) equation at screening or at baseline
* Subject has surgery scheduled to be performed without CPB ("off-pump")
* Subject has surgery scheduled for aortic dissection
* Subject is scheduled for CABG and/or valve surgery combined with additional non-emergent cardiac surgeries, e.g. for atrial fibrillation ablation
* Subject is scheduled to undergo trans catheter aortic valve implantation (TAVI) or trans catheter aortic valve replacement (TAVR), or single vessel off-pump surgeries or left ventricular device (LVAD) implantation
* Subject has a requirement for any of the following within one week prior to surgery: defibrillator or permanent pacemaker, mechanical ventilation, IABP, LVAD, other forms of mechanical circulatory support (MCS) (Note: The prophylactic insertion of an IABP preoperatively for reasons not related to existing LV pump function is not exclusionary)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-03-16 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Agervald, MD PhD, Study Director — Guard Therapeutics AB
Locations (1):
- Münster University Hospital, Münster, Germany

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: In this study, 13 subjects were enrolled, ie agreed to participate in the study following completion of the informed consent process. However, 1 subject did not fulfill all eligibility criteria and was not randomization. Hence, 12 subjects started the study, ie were assigned to one of the treatment arms.
Groups:
- RMC-035: Participants received RMC-035 intravenously
  RMC-035: Multiple dosing during 48 hours following cardiac surgery
- Placebo: Participants received matching placebo solution intravenously
  Placebo: Multiple dosing during 48 hours following cardiac surgery
Period: Overall Study
Arm/Group | RMC-035 | Placebo
Started | 8 | 4
Completed | 7 | 4
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | RMC-035 | Placebo | Total
Number analyzed (Participants) | 8 | 4 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 3
  >=65 years | 7 | 2 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.6 (8.7) | 70.4 (14.1) | 73.3 (10.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 6 | 4 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 8 | 3 | 11
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 8 | 4 | 12
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Germany | 8 | 4 | 12
Weight [Mean (Standard Deviation); unit: kilogram] | 89.75 (14.84) | 78.75 (2.99) | 86.08 (13.11)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 29.04 (3.42) | 24.99 (0.71) | 27.69 (3.40)
eGFR [Mean (Standard Deviation); unit: mL/min/1.73m^2] | 52.6 (16.5) | 76.0 (6.3) | 60.4 (17.8)

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Adverse Events (AEs)
Description: * number (%) of subjects with at least one AE
  * number (%) of subjects with at least one SAE
  * number (%) of subjects with at least one Treatment-Emergent AE (TEAE)
  * number (%) of subjects with at least one serious TEAE
  * number (%) of subjects with at least one non-serious TEAE
  * number (%) of subjects with at least one TEAE of special interest
  * number (%) of subjects with at least one TEAEs reported as related (possible/probable) to IMP
  * number (%) of subjects with at least one TEAEs leading to withdrawal of IMP
Time Frame: Baseline through day 30
Population: All subject who received any dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | RMC-035 | Placebo
Number analyzed (Participants) | 8 | 4
Participants
  Subject with at least one AE | 6 | 1
  Subject with at least one SAE | 3 | 1
  Subjects with at least one TEAE | 5 | 1
  Subjects with at least one non-serious TEAE | 5 | 1
  Subjects with at least one serious TEAE | 2 | 1
  Subjects with at least one TEAE of special interest | 0 | 0
  Subjects with at least one TEAE reported as related (possible/probable) | 0 | 0
  Subjects with at least one TEAE leading to withdrawal of IMP | 0 | 0

2. Primary Outcome: Severity of AEs
Description: - Number of TEAEs per category (mild, moderate, severe life-threatening, death)
Time Frame: Within 4 days from first dose of IMP
Population: Number of TEAEs occurring in 5 subjects on RMC-035 (N=8) and the # of TEAEs occurring in 1 subjects on placebo (N=4)
Measure: Number; unit: TEAEs
Arm/Group | RMC-035 | Placebo
Number analyzed (Participants) | 8 | 4
TEAEs
  Mild | 3 | 1
  Moderate | 5 | 2
  Severe | 3 | 2
  Life-threatening | 1 | 0
  Death | 1 | 0

3. Secondary Outcome: Maximum Observed Concentration (Cmax)
Description: Analysis of RMC-035 concentration in plasma (AUC + t1/2) after fourth infusion.
Time Frame: Blood samples taken from pre-dose and up to two hours after start of Dose 5
Population: All subjects receiving any study drug.
Measure: Mean (Standard Deviation); unit: mikrogram / milliliter
Arm/Group | RMC-035 | Placebo
Number analyzed (Participants) | 8 | 0
mikrogram / milliliter | 12.3 (4.4) |

4. Secondary Outcome: Area Under the Curve (AUC) 0-24h
Description: Analysis of RMC-035 concentrations in plasma following the fourth infusion.
Time Frame: Blood samples taken from pre-dose and up to two hours after start of Dose 5
Population: All subjects receiving RMC-035
Measure: Mean (Standard Deviation); unit: hours * microgram / milliliter
Arm/Group | RMC-035 | Placebo
Number analyzed (Participants) | 8 | 0
hours * microgram / milliliter | 38.3 (37.7) |

5. Secondary Outcome: Elimination Half-life (T1/2)
Description: Analysis of RMC-035 concentration in plasma following the fourth infusion
Time Frame: Blood samples taken from pre-dose and up to two hours after start of Dose 5
Population: All subjects receiving any RMC-035
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | RMC-035 | Placebo
Number analyzed (Participants) | 8 | 0
hours | 4.5 (1.6) |

ADVERSE EVENTS:
Time Frame: Full study period, ie baseline through day 30.
Arm/Group | RMC-035 | Placebo
All-Cause Mortality (participants affected / at risk) | 1/8 | 0/4
Serious Adverse Events (participants affected / at risk) | 3/8 | 1/4
Other Adverse Events (participants affected / at risk) | 6/8 | 1/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RMC-035 (N=8) | Placebo (N=4)
Cardiac tamponade (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 1 | 0
Anaphylactoid reaction (Infections and infestations) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0
Pneumonia (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | RMC-035 (N=8) | Placebo (N=4)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Arrhythmia supraventricular (Cardiac disorders) | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0
Small intestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Impaired healing (General disorders) | 1 | 0
Postoperative wound infection (Infections and infestations) | 1 | 1
Urinary tract infection (Infections and infestations) | 1 | 0
Hypothyroidism (Metabolism and nutrition disorders) | 1 | 0
Respiratory failure (Metabolism and nutrition disorders) | 0 | 1
Rib fracture (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-12-22): https://cdn.clinicaltrials.gov/large-docs/16/NCT04829916/Prot_003.pdf
  • Statistical Analysis Plan (2021-06-11): https://cdn.clinicaltrials.gov/large-docs/16/NCT04829916/SAP_004.pdf